CLINICAL TRIAL: NCT00889005
Title: Prevention of Post-traumatic Stress Disorder by Telephone Based Cognitive Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Aria Shalev, Professor of Psychiatry, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Shalev_Phone_2009
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-02

CONDITIONS: Stress Disorder - Post-traumatic (Acute)
Keywords: Post-traumatic Stress Disorder; Acute Stress Disorder; Cognitive behavioral therapy; Secondary Prevention; Anxiety disorders; Service Delivery
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Five sessions of trauma-focused, telephone based cognitive behavioral therapy, followed by assessment and referral to clinical treatment if needed.
  Interventions: Other: Telephone Based Cognitive Behavioral Therapy
- Waitlist control group (No Intervention): Five weeks without active intervention, followed by assessment and referral to clinical treatment if needed.

INTERVENTIONS:
Other: Telephone Based Cognitive Behavioral Therapy — Five biweekly sessions of telephone based, trauma focused cognitive behavioral therapy with homework assignment
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This is a randomized controlled study comparing telephone-based cognitive behavioral therapy (CBT) for recent survivors of traumatic events with Acute Stress Disorder (ASD) or acute PTSD with a waitlist control group. Survivors with PTSD from both groups will receive face-to-face CBT one month from the traumatic event. The study's main hypothesis is that early telephone-based CBT will reduce the prevalence of PTSD three and eight months after the traumatic event.

DETAILED DESCRIPTION:
Post-traumatic Stress Disorder (PTSD) is a prevalent and pervasive mental disorder. Studies have shown that there is a significant reluctance to use mental health services by trauma-exposed individuals at high risk for developing PTSD. Providing clinical services in combat or disaster zone might be difficult. Trauma-focused cognitive behavioral therapy (CBT) effectively reduces the prevalence of PTSD among recent survivors. Telephone based CBT was found to be effective in mood and anxiety disorders, but has not been tried in PTSD. Establishing the effectiveness of telephone based CBT has significant service delivery and public health implications. Preventing PTSD significantly reduces individuals' suffering and disability We will screen, by telephone, up to 1200 survivors of traumatic events, from a general hospital emergency department trauma registry list, randomize the first 240 with ASD or Acute PTSD to either early, telephone based cognitive behavioral therapy (ET_CBT) (n=120) or a no-treatment control condition (n=120). We will provide five sessions of ET-CBT to the former and compare the two groups three and eight months later.

Survivors from both groups who will continue to have PTSD at three months (after either treatment or waiting list), will receive 12 sessions of face-to-face, trauma focused CBT. A first phase of the study will consist of establishing the acceptance of ET-CBT and its main components (e.g., exposure to traumatic reminders) by survivors, and optimizing the protocol. It will involve 20 survivors and no randomization. Subsequent to that phase we will start recruiting for the main study. The study's main hypothesis is that early CBT will reduce the prevalence of PTSD three and eight months after the traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Exposure to psychologically traumatic events
* Diagnosis of Acute Stress Disorder or Post-traumatic Stress Disorder
* Up to four weeks after trauma exposure

Exclusion Criteria:

* Chronic PTSD
* Past and present psychosis, bipolar disorder, opiate or stimulants use
* Medical or surgical condition that interfere with subjects ability to participate in the study or sign an informed consent
* Lack of fluency in the study's main language (Hebrew)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Y Shalev, M.D., Principal Investigator — Hadassah University Hospital, Jerusalem
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control Group
Started | 65 | 74
Completed | 57 | 72
Not Completed | 8 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: Recent trauma survivors recruited following admission to a general hospital emergency room following traumatic events. Consecutive survivors screened and enrolled if eligible
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control Group | Total
Number analyzed (Participants) | 65 | 74 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.83 (12.2) | 37.95 (12.71) | 37.89 (10.4)
Sex/Gender, Customized [Number; unit: participants]
  Female | 35 | 42 | 77
  Male | 30 | 32 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 65 | 74 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 65 | 74 | 139

OUTCOME MEASURES:

1. Primary Outcome: Severity of PTSD Symptoms
Description: Clinician Administered PTSD Scale for DSM IV (CAPS IV) Score range 0-136 points Score above 40 indicate probable PTSD PTSD diagnosis inferred using DSM IV diagnostic criteria
Time Frame: Up to ten months
Population: Survivors of traumatic event with Acute PTSD symptoms one month after trauma exposure
Measure: Mean (95% Confidence Interval); unit: CAPS total Score at treatment end
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control Group
Number analyzed (Participants) | 56 | 73
CAPS total Score at treatment end | 43.4 [33.9 to 45.8] | 43.9 [41.3 to 51.6]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Waitlist Control Group; Test type: Superiority or Other; p = 0.927, ANOVA

ADVERSE EVENTS:
Arm/Group | Cognitive Behavioral Therapy | Waitlist Control Group
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/74
Other Adverse Events (participants affected / at risk) | 0/65 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No